CLINICAL TRIAL: NCT04468646
Title: To Determine the Efficacy of Neurokinin 1 Receptor Antagonist as a Therapeutic Tool Against Cytokine Storm and Respiratory Failure in Covid-19 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Fridoon Jawad Ahmad (Other)
Collaborators: University of Lahore (Other); Bahria International Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Fridoon Jawad Ahmad, Professor, head of Physiology department, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UniversityHSL-NK1R
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Neurokinin 1 Receptor, Substance P, Respiratory Illness, Inflammation, Covid-19, Coronavirus
Keywords: neurokinin 1 receptor; Substance P; Respiratory illness; inflammation; Covid-19; Coronavirus
MeSH Terms: conditions — Inflammation; COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): matching placebo drug
  Interventions: Drug: NK-1R antagonist
- NK-1R antagonist group (Experimental): 80 mg daily
  Interventions: Drug: NK-1R antagonist

INTERVENTIONS:
Drug: NK-1R antagonist — NK-1R antagonist, 80 mg daily once for 3-5 days along with dexamethasone 6 mg daily for 5 days

SUMMARY:
This is a randomized, randomized controlled trial to investigate the efficacy and safety of Neurokinin-1 Receptor (NK-1R) 80 mg orally given daily to treat cytokine storm causing inflammatory lung injury and respiratory failure associated with severe or critical COVID-19 infection. NK-1R is the receptor of Substance P (SP) and responsible for its functionality. Here, we propose that SP via its tachykinin receptor, NK-1R may cause inflammation in Covid-19 infection. It may initiate the cytokine storming via binding to its receptor NK-1 and many inflammatory mediators are released. If SP release is reduced by NK-1R antagonist, it may control the cytokine storming and hence the hyper-responsiveness of the respiratory tract through reduction in cytokine storming It may serve as the treatment strategy for Covid-19 infected patients.

Patients fulfilling the inclusion criteria will be enrolled after giving consent. They wll be randomized to treatment with either NK-1R antagonist or placebo in addition to Dexamethasone as a standard treatment given to both groups for Covid-19 infection as per the protocol at the treating hospital. Inflammatory lab markers as detailed should be collected once per day in the morning, preferably at the same time every morning. All enrolled participants will have whole blood collected for whole genome sequencing.

DETAILED DESCRIPTION:
Objective:

To evaluate the clinical outcomes of Neurokinin 1 Receptor antagonist in Covid-19 patients against the usual treatments as controls

Dosage Aprepitant capsules may be given to patients from 3-5 days fosaprepitant dimeglumine (Injection 115mg, prodrug form of aprepitant) may be substituted for oral drug in case of critical patients May be taken with or without food

Administration One capsule of Aprepitant once a day for 3-5 days

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* Both genders
* Lab Confirmed COVID-19 infection by PCR or plasma positive of specific antibody against COVID-19
* In hospital treatment ≥ 72 hours
* Admitted patients
* Severe Disease (Respiratory rate >=30/min; or (b) Rest SPO2<=90%; or (c) PaO2/FiO2<=300 mmHg) or
* Critical Phase (Respiratory failure and needs mechanical ventilation; or Shock occurs; or Multiple organ failure and needs ICU monitoring)

Exclusion Criteria:

* Patients who are not willing to give consent
* known HIV,HBV, HCV infection
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to improvement on a 7-point ordinal scale as compared to baseline | 14 days or discharge

SECONDARY OUTCOMES:
total in-hospital days and the total duration | 14 days or discharge
Treatment and prevention of inflammatory lung injury as measured by change in baseline of interleukin-6 (IL-6) | 14 days or discharge
Rate of Decline of COVID-19 viral load assessed by RT-PCR from nasopharyngeal samples | 14 days or discharge
Reduction from baseline of NRS for cough | 14 days or discharge
Reduction from baseline of NRS for nausea | 14 days or discharge
Time to normalization of fever for at least 48 hours | 14 days or discharge
Time to improvement in oxygenation for at least 48 hours | 14 days or discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria International Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No